CLINICAL TRIAL: NCT04791852
Title: Potential Role of Donor-derived Cell-Free DNA as a Biomarker in Cardiac Allograft Vasculopathy
Acronym: FreeDNA-CAV
Status: Completed | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Javier Segovia Cubero, Head of Cardiology Department, Puerta de Hierro University Hospital
Other Study IDs: FreeDNA-CAV
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Donor-derived Cell Free DNA; Heart Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Donor-derived Cell Free DNA — We will compare ddcfDNA with coronary angiogram determined CAV grading, according to ISHTL2010 classification

SUMMARY:
Cross-sectional study. We will prospectively obtain ddcf-DNA levels in all patients who undergo routine coronary angiography > 1 year after HT. Our main goal is to evaluate the performance of Donor-derived Cell Free DNA (ddcf-DNA) as a biomarker of CAV.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 80 years old, HT > 1 year ago

Exclusion Criteria:

* Patients under 18 or over 80 years old
* Multiorgan transplant
* History of acute cellular rejection ≥ 1R or antibody mediated rejection in the previous 6 months
* Concomitant infection by CMV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant recipients that undergo routine surveillance coronary angiogram
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Correlation between ddcf-DNA and CAV | 2 years
  Correlation between ddcf-DNA levels and the presence of any degree of CAV (CAV0 vs CAV1, 2, or 3)
Performance of the biomarker for the diagnosis of CAV | 2 years
  Determine the performance of this biomarker in this situation using receiver-operator characteristics analysis.

SECONDARY OUTCOMES:
Correlation of ddcf-DNA with the different degrees of CAV (0, 1, 2 and 3) | 2 years
  Correlation of ddcf-DNA with the different degrees of CAV (0, 1, 2 and 3)
Correlation of ddcf-DNA with other biomarkers (NTproBNP and troponin I) | 2 years
  Correlation of ddcf-DNA with other biomarkers (NTproBNP and troponin I)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jimenez-Blanco Bravo M, Perez-Gomez L, Hernandez-Perez FJ, Arellano-Serrano C, Torres-Sanabria M, Gomez-Bueno M, Oteo-Dominguez JF, Mingo-Santos S, Segovia-Cubero J. Lack of Usefulness of Donor-Derived Cell-Free DNA as a Biomarker for Cardiac Allograft Vasculopathy: A Prospective Study. Front Cardiovasc Med. 2022 Apr 6;9:856600. doi: 10.3389/fcvm.2022.856600. eCollection 2022. PMID 35463750